CLINICAL TRIAL: NCT05351970
Title: Barbed Suture vs. Monofilament for Emergency Midline Laparotomy Closure, a Retrospective Analysis
Brief Title: Barbed Suture for Emergency Midline Laparotomy Closure
Acronym: BAROTOMY
Status: Completed | Type: Observational
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, Luis Sánchez Guillen, Clinical Professor Luis Sánchez-Guillén, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Other Study IDs: BAROTOMY
Record Dates: First submitted 2022-04-18; First posted 2022-04-28 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Incisional Hernia of Midline of Abdomen
Keywords: incisional hernia; midline laparotomy; urgency laparotomy; barbed suture; monofilament suture
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Monofilament closure: Patients with midline emergency laparotomy, which closure was performed with monofilament suture
- Barbed closure: Patients with midline emergency laparotomy, which closure was performed with barbed suture
  Interventions: Procedure: Barbed

INTERVENTIONS:
Procedure: Barbed — Efficacy of barbed and monofilament closure regarding incisional hernia
  Groups: Barbed closure

SUMMARY:
Urgency surgeries are often performed in a stressful setting with critical patient involved. In this context, laparotomy closure can sometimes be the most neglected part of the procedure. Barbed sutures, frequently used in laparoscopic procedures, have proven to be effective in maintaining traction.

The aim of this study is to describe the incisional hernia rate after emergency midline laparotomy, according to the suture utilized, evaluated at one month and one year postoperative.

DETAILED DESCRIPTION:
A retrospective cohort study was performed including patients with urgency midline laparotomy during 2018-2019. Group A was represented by patients with slowly absorbable monofilament continuous suture, while Group B included patients with barbed suture closure.

Main variables were hernia rates one month and one year after surgery, diagnosed by physical exploration and/or imaging. Demographic characteristics, risk factors, among other descriptive determinations were registered.

A total of 128 patients were performed an emergency midline laparotomies, and 110 meet all inclusion criteria. There was equality between sex and median age was 65 years old. Significative differences were observed regarding incisional hernia at 30 days, being less frequent when barbed suture was utilized. These differences were not present at the long-term reevaluation (one year).

In conclusion, midline laparotomy closure must be performed within quality standards. The lack of studies regarding emergency laparotomy closure, the European Hernia Society stated that no recommendations can be given on this patients. Barbed suture appears as a promising option for closure in these specific circumstances, but needs further study.

ELIGIBILITY:
Inclusion Criteria:

* Emergency laparotomy
* Minimum age of 18 years old.
* Digestive surgical disease.
* Minimum survival of one month postoperatively.

Exclusion Criteria:

* Laparoscopic surgical procedure.
* Non-digestive surgical procedure (gynecology, urology...).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with emergency laparotomy performed due to digestive surgical disease.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Incisional Hernia 1 month | Hernia 1 month
  Incidence of incisional hernia at one month after surgery
Incisional Hernia 1 year | Hernia 1 year
  Incidence of incisional hernia at one year after surgery

SECONDARY OUTCOMES:
Surgical Site Infection | 1 month
  Incidence of postoperative surgical site infection
Evisceration | 1 month
  Incidence of early abdominal evisceration
Medical complications | 1 month
  Incidence of other medical complications

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Universitario de Elche, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Israelsson LA, Millbourn D. Prevention of incisional hernias: how to close a midline incision. Surg Clin North Am. 2013 Oct;93(5):1027-40. doi: 10.1016/j.suc.2013.06.009. PMID 24035074
- [Background] NELA (National Emergency Laparotomy Audit). Seventh Patient Report of the National Emergency Laparotomy Audit. December 2019 - November 2020.
- [Background] Diener MK, Voss S, Jensen K, Buchler MW, Seiler CM. Elective midline laparotomy closure: the INLINE systematic review and meta-analysis. Ann Surg. 2010 May;251(5):843-56. doi: 10.1097/SLA.0b013e3181d973e4. PMID 20395846
- [Background] Muysoms FE, Antoniou SA, Bury K, Campanelli G, Conze J, Cuccurullo D, de Beaux AC, Deerenberg EB, East B, Fortelny RH, Gillion JF, Henriksen NA, Israelsson L, Jairam A, Janes A, Jeekel J, Lopez-Cano M, Miserez M, Morales-Conde S, Sanders DL, Simons MP, Smietanski M, Venclauskas L, Berrevoet F; European Hernia Society. European Hernia Society guidelines on the closure of abdominal wall incisions. Hernia. 2015 Feb;19(1):1-24. doi: 10.1007/s10029-014-1342-5. Epub 2015 Jan 25. PMID 25618025
- [Background] Peden CJ, Aggarwal G, Aitken RJ, Anderson ID, Bang Foss N, Cooper Z, Dhesi JK, French WB, Grant MC, Hammarqvist F, Hare SP, Havens JM, Holena DN, Hubner M, Kim JS, Lees NP, Ljungqvist O, Lobo DN, Mohseni S, Ordonez CA, Quiney N, Urman RD, Wick E, Wu CL, Young-Fadok T, Scott M. Guidelines for Perioperative Care for Emergency Laparotomy Enhanced Recovery After Surgery (ERAS) Society Recommendations: Part 1-Preoperative: Diagnosis, Rapid Assessment and Optimization. World J Surg. 2021 May;45(5):1272-1290. doi: 10.1007/s00268-021-05994-9. Epub 2021 Mar 6. PMID 33677649
- [Background] Velotti N, Manigrasso M, Di Lauro K, Vertaldi S, Anoldo P, Vitiello A, Milone F, Musella M, De Palma GD, Milone M. Barbed suture in gastro-intestinal surgery: A review with a meta-analysis. Surgeon. 2022 Apr;20(2):115-122. doi: 10.1016/j.surge.2021.02.011. Epub 2021 Apr 2. PMID 33820730
- [Background] Angioli R, Plotti F, Montera R, Damiani P, Terranova C, Oronzi I, Luvero D, Scaletta G, Muzii L, Panici PB. A new type of absorbable barbed suture for use in laparoscopic myomectomy. Int J Gynaecol Obstet. 2012 Jun;117(3):220-3. doi: 10.1016/j.ijgo.2011.12.023. Epub 2012 Mar 23. PMID 22445426
- [Background] Sundaram K, Piuzzi NS, Klika AK, Molloy RM, Higuera-Rueda CA, Krebs VE, Mont MA. Barbed sutures reduce arthrotomy closure duration and suture utilisation compared to interrupted conventional sutures for primary total hip arthroplasty: a randomised controlled trial. Hip Int. 2021 Sep;31(5):582-588. doi: 10.1177/1120700020911891. Epub 2020 Mar 19. PMID 32188284
- [Background] Lin YF, Lai SK, Liu QY, Liao BH, Huang J, Du L, Wang KJ, Li H. Efficacy and safety of barbed suture in minimally invasive radical prostatectomy: A systematic review and meta-analysis. Kaohsiung J Med Sci. 2017 Mar;33(3):107-115. doi: 10.1016/j.kjms.2016.12.005. Epub 2017 Jan 27. PMID 28254112
- [Background] Mingoli A, Puggioni A, Sgarzini G, Luciani G, Corzani F, Ciccarone F, Baldassarre E, Modini C. Incidence of incisional hernia following emergency abdominal surgery. Ital J Gastroenterol Hepatol. 1999 Aug-Sep;31(6):449-53. PMID 10575560
- [Background] National Healthcare Safety Network (NHSN). Surgical Site Infection. Jan 2022;39,11.
- [Background] Morales S, Barreriro F, Hernández P, Feliu X. Cirugía de la pared abdominal. Asocación Española de Cirujanos; 2º Ed; Madrid; 2013: Sección III y VI.
- [Background] Ruiz-Tovar J, Llavero C, Jimenez-Fuertes M, Duran M, Perez-Lopez M, Garcia-Marin A. Incisional Surgical Site Infection after Abdominal Fascial Closure with Triclosan-Coated Barbed Suture vs Triclosan-Coated Polydioxanone Loop Suture vs Polydioxanone Loop Suture in Emergent Abdominal Surgery: A Randomized Clinical Trial. J Am Coll Surg. 2020 May;230(5):766-774. doi: 10.1016/j.jamcollsurg.2020.02.031. Epub 2020 Feb 27. PMID 32113031
- [Background] Clapp B, Klingsporn W, Lodeiro C, Wicker E, Christensen L, Jones R, Tyroch A. Small bowel obstructions following the use of barbed suture: a review of the literature and analysis of the MAUDE database. Surg Endosc. 2020 Mar;34(3):1261-1269. doi: 10.1007/s00464-019-06890-z. Epub 2019 Jun 10. PMID 31183792
- [Background] Rahbari NN, Knebel P, Kieser M, Bruckner T, Bartsch DK, Friess H, Mihaljevic AL, Stern J, Diener MK, Voss S, Rossion I, Buchler MW, Seiler CM. Design and current status of CONTINT: continuous versus interrupted abdominal wall closure after emergency midline laparotomy - a randomized controlled multicenter trial [NCT00544583]. Trials. 2012 May 30;13:72. doi: 10.1186/1745-6215-13-72. PMID 22647387
- See also: Johnson-Johnson catalogue — https://emeatotalaccess.showpad.com/share/5a4JwkPiLJ0o8alBcXV7G/0